CLINICAL TRIAL: NCT03352765
Title: A Phase I Study of Bendamustine and Melphalan Conditioning and Autologous Stem Cell Transplantation for Treatment of Multiple Myeloma and Relapsed/Refractory B-cell Lymphoma in Elderly Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-373
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma
Keywords: Rituximab; Bendamustine; Melphalan; Autologous Stem Cell Transplantation (ASCT); 17-373
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Bendamustine Hydrochloride; Melphalan

STUDY DESIGN:
Intervention Model Description: This is a phase I single arm, open label trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- rituximab, bendamustine & melphalan and ASCT (Experimental): This is a phase I study of rituximab, bendamustine and melphalan (RBM) conditioning followed by ASCT in elderly patients with B-cell NHL. Conditioning regimen consist of rituximab 375 mg/m2 on days -11 and -4, bendamustine 160 mg/m2 intravenously on days -3 and -2; melphalan 140 mg/m2 intravenously on day -1 before the reinfusion of autologous stem cells on day 0. The conditioning timeline can be modified if there are patient scheduling conflicts. Patients who are deemed inevaluable will be replaced for the primary objective. Patients will be considered inevaluable if they don't receive one dose of conditioning regimen and are removed from the study.
  Interventions: Drug: rituximab; Drug: bendamustine; Drug: melphalan; Procedure: Autologous Stem Cell Transplantation (ASCT)

INTERVENTIONS:
Drug: rituximab — rituximab 375 mg/m2 on days -11 and -4, The second dose of rituximab (day -4) is administered 7 days after the first dose (day -11), +/- 1 day. Rituximab may be administered by a local oncologist. If the participant has a CD20 negative tumor, rituximab can be omitted from the conditioning regimen.
Drug: bendamustine — bendamustine 160 mg/m2 intravenously on days -3 and -2
Drug: melphalan — melphalan 140 mg/m2 intravenously on day -1 before the reinfusion of autologous stem cells on day 0.
Procedure: Autologous Stem Cell Transplantation (ASCT) — reinfusion of autologous stem cells on day 0.

SUMMARY:
This study is testing a combination of chemo-immuno therapy called RBM. RBM consists of combination of drugs: rituximab, bendamustine, and melphalan followed by reinfusion of the participants own stem cells which is called autologous stem cell transplant (ASCT). Compared to the standard BEAM regimen, this RBM regimen may or may not be less effective in lymphoma, but will likely have fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

Phase I eligibility:

* Any patient with multiple myeloma B-cell non-Hodgkin lymphoma would be eligible for phase I portion of the study.

Dose expansion eligibility:

* Histologically confirmed diagnosis of multiple myeloma or rel/ref DLBCL, or diffuse large B cell lymphoma transformed from an indolent lymphoma Since the endpoint of the Phase I portion is safety, any patient with myeloma or B-cell NHL can be enrolled. For dose expansion study patients with myeloma and B-NHL will be analyzed separately. The PFS endpoint varies greatly amongst different types of lymphoma. In order to accurately interpret the survival data as secondary endpoint, a homogeneous cohort of patients with DLBCL will be evaluated. DLBCL is the most aggressive B-NHL with limited options. Other B-NHL's are generally more indolent and have more options available to them.

Additional eligibility for both the phase I and dose expansion cohort:

* Patients between the ages of 65 to 69 years old with a Hematopoietic Stem Cell Transplant Comorbidity Index (HCT-CI) score of 3 or higher.
* Any patient age 70 years old or older, irrespective of their Hematopoietic Stem Cell Transplant Comorbidity Index (HCT-CI) score.
* KPS ≥ 70
* Males must agree to use an acceptable form of contraception per institutional practices.
* Complete or partial response to salvage chemotherapy by IWG Working Group Criteria
* Cardiac ejection fraction of ≥ 45%
* Hemoglobin-adjusted diffusing capacity of carbon monoxide (DLCO) of ≥45%
* Creatinine clearance of ≥50 mL/min
* Completion of most recent salvage therapy within 8 weeks of enrollment
* Direct bilirubin ≤2.0 mg/dL in the absence of suspected Gilbert's disease (if Gilbert's disease is suspected, the total bilirubin must be ≤3.0 mg/dL), and AST ≤ 2.5 ULN.

Exclusion Criteria:

* In Lymphoma: Disease progression by IWG Working Group Criteria since last therapy
* Patients with history of CNS involvement
* Prior autologous (only in lymphoma) or allogeneic stem cell transplantation
* Patients who have failed bendamustine-based regimen previously
* Patients within 6 months of MI and stroke will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | 1 year
  are defined as grade > 3, non-hematologic toxicity related to treatment excluding grade 3 nausea or vomiting responsive to anti-emetic treatment, grade 3 diarrhea responding to anti-diarrheal treatment, grade 3 fatigue, grade 3 skin rash responsive to topical or systemic steroids, grade 3 fevers (> 40 degrees Celsius for < 24 hours) and alopecia per CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Parastoo Dahi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/